CLINICAL TRIAL: NCT00650845
Title: Renal Safety Evaluation After Dotarem®-Enhanced MRI Compared With Non-enhanced MRI in Patients at High Risk of Developing Contrast Medium Induced Nephropathy
Brief Title: Renal Safety Evaluation After Dotarem®-Enhanced MRI
Acronym: RESCUE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DGD-44-044
Record Dates: First submitted 2008-03-04; First posted 2008-04-02 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-03

CONDITIONS: Renal Insufficiency
Keywords: contrast-induced nephropathy, creatinemia
MeSH Terms: conditions — Renal Insufficiency | interventions — gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dotarem®-enhanced MRI (Experimental): Patients undergoing Dotarem®-enhanced MRI for diagnostic purposes
  Interventions: Drug: Dotarem®-enhanced MRI
- Non-enhanced MRI (Other): Patients undergoing non-enhanced MRI for diagnostic purposes
  Interventions: Other: non-enhanced MRI

INTERVENTIONS:
Drug: Dotarem®-enhanced MRI — Single IV administration before MRI exam
  Other Names: Gadoterate meglumine; Gadoteric acid
  Arms: Dotarem®-enhanced MRI
Other: non-enhanced MRI — non injected MRI
  Other Names: unenhanced MRI
  Arms: Non-enhanced MRI

SUMMARY:
Although there is a well documented risk of acute renal failure with the iodinated contrast agents, the implication of intravenous gadolinium-based contrast agents in nephrotoxicity remains controversial. The aim of this study was to evaluate the safety profile of gadoterate meglumine (Dotarem®) in patients with chronic renal insufficiency by evaluating the rate of patients experiencing contrast-induced nephrotoxicity following the injection of gadoterate meglumine.

DETAILED DESCRIPTION:
Patients with renal insufficiency not requiring hemodialysis and scheduled to undergo a contrast enhanced MRI or unenhanced MRI examination to specify a diagnosis, were selected for inclusion. Two groups of patients were defined on the basis of the planned imaging procedure selected to obtain a diagnosis: those undergoing a Dotarem®-enhanced MRI and those undergoing an unenhanced MRI.

A clinically significant increase in serum creatinine levels after the contrast-enhanced MRI exam was used as an indication of contrast induced nephrotoxicity. A blood test was performed 24h before the MRI in order to evaluate baseline creatinine values. 72h after the exam, a second blood test was performed. An increase in creatinemia above 25% from baseline levels was defined as a contrast-induced nephrotoxic reaction. The primary endpoint of the study assessed the percentage of patients presenting a contrast-induced nephrotoxic reaction in order to show a non inferiority of enhanced as compared to non-enhanced MRI exams.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, > or equal 18 years ;
* Patient with a known stable renal insufficiency ;
* Patient scheduled to undergo an MRI examination to specify a diagnosis ;
* Patient able to understand and provide written informed consent to participate in the trial ;

Exclusion Criteria:

* Patient with a contra-indication to MRI ;
* Patient who has a diagnosis of an hemodynamic instability or acute myocardial infarction within 15 days prior the inclusion ;
* Patient who needs hemodialysis ;
* Patient with known allergy to gadolinium chelates ;
* Patient receiving medications known to be nephrotoxic or to cause increases in serum creatinine level within 2 weeks before the inclusion ;
* Patients planned to either undergo surgery or receive chemotherapy ;
* Any condition which, based on the investigator's clinical judgement, would prevent the patient from completing all trial assessments and visits ;
* Patient under guardianship and/or inability or unwillingness to cooperate with the requirements of this trial ;
* Patient with newly discovered unstable diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2008-01; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Deray, Pr, MD, PhD, Principal Investigator — Groupe Hospitalier Pitie-Salpetriere
Locations (15):
- Belgium (3):
  - Onze Lievevrouwziekenhuis, Aalst
  - University Hospital Ghent, Ghent
  - Alg. Inwendige Ziekten -Nierziekten, Roeselare
- France (8):
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Hôpital A. Calmette, Lille
  - Hôpital Edouard Herriot, Lyon
  - Hopital Pitie Salpetriere, Paris
  - Hopital Bichat, Paris
  - Hôpital Tenon, Paris
  - CHU Strasbourg, Strasbourg
  - Hôpital Trousseau, Tours
- Italy (2):
  - Azienda Ospedaliera Universitaria di Ferrara, Ferrara
  - Ente Ospedaliero Ospedali Galliera,, Genova
- Spain (2):
  - Hospital San Carlos, Madrid
  - Hospital Dr PESET, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study did not use randomization. Eligible patients who provided written consent were enrolled chronologically in each investigational center. A total of 142 patients were screened between 29 January 2008 and 05 May 2011, 135 of whom were included in 15 European centers, eight centers in France, three in Belgium, two in Spain and two in Italy.
Pre-assignment Details: 10 patients were screened but did not undergo the planned procedure: 7 were screen failures and 3 were included but dropped out prior to undergoing the planned procedure. Hence the total number of patients who were assigned to both groups is 132.
Groups:
- Dotarem®-Enhanced MRI: Dotarem®: Single IV administration
Period: Overall Study
Arm/Group | Dotarem®-Enhanced MRI | Non-enhanced MRI
Started | 75 | 57
Completed | 70 | 44
Not Completed | 5 | 13
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Protocol Violation | 0 | 13

BASELINE CHARACTERISTICS:
Groups:
- Dotarem®-Enhanced MRI: Dotarem®: Single IV administration before the MRI
- Total: Total of all reporting groups
Arm/Group | Dotarem®-Enhanced MRI | Non-enhanced MRI | Total
Number analyzed (Participants) | 75 | 57 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (11.5) | 66.2 (12.2) | 67.9 (12.0)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 20 | 44
  >=65 years | 51 | 37 | 88
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 51 | 34 | 85
Region of Enrollment [Number; unit: participants]
  France | 44 | 11 | 55
  Belgium | 14 | 7 | 21
  Spain | 17 | 23 | 40
  Italy | 0 | 16 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Presenting Contrast-induced Nephropathy as Defined by an Increase in Serum Creatinine Levels of a Least 25% Over Baseline Levels, in the Full Analysis Set Population.
Description: Comparing the number of patients experiencing an increase of creatinine of at least 25% over baseline levels after Dotarem®-enhanced MRI and after non-enhanced MRI in patients with at least a moderate renal insufficiency.
Time Frame: baseline pre MRI and 3 days post MRI
Population: Full analysis set population: all included patients with a pre and post-procedure blood sample for creatinine measures.
Measure: Number; unit: Number of patients
Arm/Group | Dotarem®-Enhanced MRI | Non-enhanced MRI
Number analyzed (Participants) | 70 | 44
Number of patients | 1 | 0
Statistical Analysis 1: Comparison: Dotarem®-Enhanced MRI vs Non-enhanced MRI; The clinical non-inferiority limit of (non-enhanced - Dotarem®-enhanced) was fixed at -15%. The exact 95%Confidence Interval (CI) of the difference (non-enhanced - Dotarem®-enhanced) was [-7.9%; +6.7%]; Test type: Non-Inferiority or Equivalence — Assuming that in both MRI groups approximately 12% of the patients would have an increase in serum creatinine of at least 25% with respect to baseline values after imaging procedures, 120 evaluable patients (2 x 60) were needed to ensure with 80% power, at 5% one-sided significance level, that the difference between the two MRI procedures was less than 15% which was the non-inferiority clinical limit of the difference established for this study; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-7.9 to 6.7]

2. Secondary Outcome: Percent Change of Serum Creatinine Level From Baseline to 72±24 Hours After Examination, in the Full Analysis Set Population.
Description: Serum creatinine levels were measured at baseline and at 72±24 hours after examination. The percentage of change in creatinemia from baseline was calculated for both the Dotarem® and the non-enhanced groups.
Time Frame: Baseline pre MRI and 3 days post MRI
Population: Full analysis set population:all included patients with a pre and post-procedure blood sample for creatinine measurement.
Measure: Mean (Standard Deviation); unit: Percentage of change from baseline
Arm/Group | Dotarem®-Enhanced MRI | Non-enhanced MRI
Number analyzed (Participants) | 70 | 44
Percentage of change from baseline | -1.40 (10.36) | -3.48 (9.92)
Statistical Analysis 1: Comparison: Dotarem®-Enhanced MRI vs Non-enhanced MRI; Serum creatinine level fluctuation in terms of difference between baseline and 72 ±24hours after imaging procedure values was computed for both MRI procedures and compared between the 2 groups. A linear regression model was used to model the serum creatinine changes from baseline as a function of the MRI procedure with adjustment on centers; Test type: Superiority or Other; p = 0.291, t-test, 2 sided — p-value for main effect (difference between groups) adjusted on centers

3. Primary Outcome: Number of Patients Presenting Contrast-induced Nephropathy as Defined by an Increase in Serum Creatinine Levels of at Least 25% Over Baseline Levels, in the Per Protocol Population.
Description: as for outcome 1
Time Frame: Baseline pre MRI and 3 days post MRI
Population: Per protocol population: This population is comprised of the full analysis set population (i.e. all included patients with a pre and post-procedure blood sample for creatinine measurement) deprived of patients with protocol deviations/violations.
Measure: Number; unit: Number of patients
Arm/Group | Dotarem®-Enhanced MRI | Non-enhanced MRI
Number analyzed (Participants) | 37 | 30
Number of patients | 1 | 0
Statistical Analysis 1: Comparison: Dotarem®-Enhanced MRI vs Non-enhanced MRI; The clinical non-inferiority limit of (non-enhanced - Dotarem®-enhanced) was fixed at -15%. The exact 95%CI of the difference (non-enhanced - Dotarem®-enhanced) was [-14.1%; +8.9%]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-14.1 to 8.9]

4. Secondary Outcome: Percent Change of Serum Creatinine Level Variation From Baseline to 72±24 Hours After Examination, in the Per Protocol Population
Description: as for outcome 2
Time Frame: Baseline pre MRI and 3 days post MRI
Population: Per protocol population. This population is comprised of the full analysis set population (i.e. all included patients with a pre and post-procedure blood sample for creatinine measurement) deprived of patients with protocol deviations/violations.
Measure: Mean (Standard Deviation); unit: Percentage of change from baseline
Arm/Group | Dotarem®-Enhanced MRI | Non-enhanced MRI
Number analyzed (Participants) | 37 | 30
Percentage of change from baseline | 0.05 (10.84) | -5.17 (9.16)
Statistical Analysis 1: Comparison: Dotarem®-Enhanced MRI vs Non-enhanced MRI; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.040, t-test, 2 sided — p-value for main effect (difference between groups) adjusted on centers

5. Secondary Outcome: Percent Change of Estimated Glomerular Filtration Rate (eGFR) Values From Baseline to 72±24 Hours After Examination, in the Full Analysis Set Population
Description: eGFR was assessed using creatinemia and the Modification of Diet in Renal Disease (MDRD) study equation. eGFR were evaluated in terms of mean difference between the pre- and post-MRI procedure. The eGFR variation was expressed as a percentage of change from baseline values.
Time Frame: Baseline pre MRI and 3 days post MRI
Population: Full analysis set population: all included patients with a pre and a post-procedure blood sample for creatinine measurements.
Measure: Mean (Standard Deviation); unit: Percentage of change from baseline
Arm/Group | Dotarem®-Enhanced MRI | Non-enhanced MRI
Number analyzed (Participants) | 70 | 44
Percentage of change from baseline | 3.02 (12.51) | 5.55 (12.94)
Statistical Analysis 1: Comparison: Dotarem®-Enhanced MRI vs Non-enhanced MRI; eGFR fluctuation in terms of percentage and mean difference between baseline and 72 ±24hours after imaging procedure values was computed for both MRI procedures and compared between the 2 groups. A linear regression model was used to model the relative or absolute eGFR variation from baseline as a function of the MRI procedure with adjustment on centers; Test type: Superiority or Other; p = 0.301, t-test, 2 sided — p-value for main effect (difference between groups) adjusted on centers

6. Secondary Outcome: eGFR Values Variation Between Baseline and 72±24 Hours After Examination, in the Per Protocol Population
Description: eGFR (estimated Glomerular Filtration Rate) was assessed using creatinemia and the Modification of Diet in Renal Disease (MDRD) study equation. eGFR were evaluated in terms of mean difference between the pre- and post-MRI procedure. The eGFR variation was expressed as a percentage of change from baseline values.
Time Frame: Baseline pre MRI and 3 days post MRI
Population: Per protocol population: This population is comprised of the full analysis set population (i.e. all included patients with a pre and a post- procedure blood sample for creatinine measurements) deprived of patients with protocol deviations/violations.
Measure: Mean (Standard Deviation); unit: Percentage of change from baseline
Arm/Group | Dotarem®-Enhanced MRI | Non-enhanced MRI
Number analyzed (Participants) | 37 | 30
Percentage of change from baseline | 1.37 (12.65) | 7.58 (12.82)
Statistical Analysis 1: Comparison: Dotarem®-Enhanced MRI vs Non-enhanced MRI; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.051, t-test, 2 sided — p-value for main effect (difference between groups) adjusted on centers

ADVERSE EVENTS:
Time Frame: The period of observation for Adverse Events (AEs) collection extended from the time of patient informed consent until the end of his/her follow-up (i.e. 72 ±24hrs or 14 days after the imaging procedure) or until patient early withdrawal from the trial.
Arm/Group | Dotarem®-Enhanced MRI | Non-enhanced MRI
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/44
Other Adverse Events (participants affected / at risk) | 6/70 | 0/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dotarem®-Enhanced MRI (N=70) | Non-enhanced MRI (N=44)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) — This adverse event was deemed not related to the injection of Dotarem®
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) — This adverse event was deemed not related to the injection of Dotarem®
Hypotension (Vascular disorders) | 1 (1) | 0 (0) — This adverse event was deemed not related to the injection of Dotarem®
Blood creatinin increased (Investigations) | 1 (1) | 0 (0) — This adverse event was deemed possibly related to the injection of Dotarem®
toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) — This adverse event was deemed not related to the injection of Dotarem®
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — This adverse event was deemed not related to the injection of Dotarem®

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished data given to the investigator may be transmitted to a third party without prior approval of the sponsor in writing. The data are the exclusive property of Guerbet.

The investigator undertakes to submit to Guerbet any draft articles or papers related to this study within 30 days of their submission to the scientific review or the congress scientific committee.

All written or oral papers and publications must have the joint agreement of the investigator and the sponsor.